CLINICAL TRIAL: NCT02986828
Title: The Long-term Effect of Platelet Rich Plasma and Hydrodissection for Patients With Carpal Tunnel Syndrome
Brief Title: Platelet Rich Plasma and Hydrodissection for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP and hydrodissection
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: platelet rich plasma; Hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Saline Solution; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet rich plasma injection (Experimental): The platelet rich plasma (PRP) is a new and potential treatment for peripheral neuropathy in many animal studies.
  Interventions: Drug: platelet rich plasma; Device: Ultrasound
- Normal saline (Active Comparator): Normal saline for ultrasound-guided hydrodissection
  Interventions: Drug: Normal saline; Device: Ultrasound

INTERVENTIONS:
Drug: platelet rich plasma — Ultrasound-guided 3cc PRP injection between proximal carpal tunnel and median nerve.
  Arms: platelet rich plasma injection
Drug: Normal saline — Ultrasound-guided 3cc normal saline injection between proximal carpal tunnel and median nerve.
  Arms: Normal saline
Device: Ultrasound

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration. The platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders and recent reports showed being beneficial for peripheral neuropathy in animal studies. Since 2014, three small clinical trials showed the positive effect of PRP in peripheral neuropathy included CTSin a pilot research. However, these studies have not entirely proved the effects of PRP on peripheral neuropathy because these studies enrolled small number of patients and lacked controlled design. The investigators design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided PRP injection in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients with bilateral CTS will been randomized into intervention and control side. Participants in intervention group received one-dose ultrasound-guided PRP injection and control side received one-dose ultrasound-guided normal saline injection. No additional treatment after injection through the study period. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 3rd, 6th month and one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 3rd, 6th month and 1 year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and 1 year after injection
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 3rd, 6th month and 1 year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and 1 year after injection
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the severity of symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 3rd, 6th month and 1 year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and 1 year after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 3rd, 6th month and 1 year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and 1 year after injection
  antidromic sensory nerve conduction velocity of the median nerve before treatment and multiple time frame after treatment.
Change from finger pinch on 2nd week, 1st, 3rd, 6th month and 1 year after injection | Pre-treatment, 2nd week, 1st, 3rd, 6th month and 1 year after injection
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Anjayani S, Wirohadidjojo YW, Adam AM, Suwandi D, Seweng A, Amiruddin MD. Sensory improvement of leprosy peripheral neuropathy in patients treated with perineural injection of platelet-rich plasma. Int J Dermatol. 2014 Jan;53(1):109-13. doi: 10.1111/ijd.12162. Epub 2013 Oct 29. PMID 24168291
- [Result] Sanchez M, Yoshioka T, Ortega M, Delgado D, Anitua E. Ultrasound-guided platelet-rich plasma injections for the treatment of common peroneal nerve palsy associated with multiple ligament injuries of the knee. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1084-9. doi: 10.1007/s00167-013-2479-y. Epub 2013 Mar 22. PMID 23519544
- [Result] Scala M, Mereu P, Spagnolo F, Massa M, Barla A, Mosci S, Forno G, Ingenito A, Strada P. The use of platelet-rich plasma gel in patients with mixed tumour undergoing superficial parotidectomy: a randomized study. In Vivo. 2014 Jan-Feb;28(1):121-4. PMID 24425846
- [Result] Malahias MA, Johnson EO, Babis GC, Nikolaou VS. Single injection of platelet-rich plasma as a novel treatment of carpal tunnel syndrome. Neural Regen Res. 2015 Nov;10(11):1856-9. doi: 10.4103/1673-5374.165322. PMID 26807124